CLINICAL TRIAL: NCT01286740
Title: A Phase 2B Open Label Pilot Study to Evaluate Switching From a Regimen Consisting of a Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF) Single Tablet Regimen (STR) to Emtricitabine/Rilpivirine/Tenofovir Disoproxil Fumarate (FTC/RPV/TDF) STR in Virologically Suppressed, HIV 1 Infected Subjects
Brief Title: Study to Evaluate Switching From a Regimen Consisting of the Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate Single-Tablet Regimen (STR) to the Emtricitabine/Rilpivirine/Tenofovir Disoproxil Fumarate STR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-264-0111
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; HIV; Treatment Experienced
MeSH Terms: interventions — Emtricitabine, Rilpivirine, Tenofovir Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FTC/RPV/TDF (Experimental): Participants switched from their existing treatment regimen of EFV/FTC/TDF to the FTC/RPV/TDF STR.
  Interventions: Drug: FTC/RPV/TDF

INTERVENTIONS:
Drug: FTC/RPV/TDF — Emtricitabine (FTC) 200 mg/rilpivirine (RPV) 25 mg/tenofovir disoproxil fumarate (tenofovir DF; TDF) 300 mg single-tablet regimen (STR) administered orally with a meal once daily
  Other Names: Complera; Eviplera

SUMMARY:
The purpose of this Phase 2b study was to evaluate the efficacy and safety of the emtricitabine/rilpivirine/tenofovir disoproxil fumarate (FTC/RPV/TDF) STR, after switching from the efavirenz (EFV)/FTC/TDF STR at baseline, in maintaining HIV-1 RNA < 50 copies/mL at Week 12. HIV-infected patients were enrolled if they had received EFV/FTC/TDF for ≥ 3 months prior to study start, were experiencing safety or tolerability concerns (in particular, EFV-related intolerance), and wished to change to an alternate, better-tolerated regimen.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* Receiving EFV/FTC/TDF continuously for ≥ 3 months preceding the screening visit
* Plasma HIV-1 RNA concentrations (at least two measurements) at undetectable levels for ≥ 8 weeks prior to the screening visit and HIV-1 RNA < 50 copies/mL at the screening visit
* On their first antiretroviral drug regimen, and no HIV-1 RNA > 50 copies/mL measured at two consecutive time points after first achieving HIV RNA < 50 copies/mL
* Had a genotype prior to starting FTC/RPV/TDF and no known resistance to any of the study agents
* Normal ECG
* Hepatic transaminases (AST and ALT) ≤ 5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm^3; platelets ≥ 50,000/mm^3; hemoglobin ≥ 8.5 g/dL)
* Serum amylase ≤ 5 x ULN (subjects with serum amylase > 5 x ULN eligible if serum lipase ≤ 5 x ULN)
* Adequate renal function (estimated glomerular filtration rate ≥ 50 mL/min according to the Cockcroft-Gault formula)
* Males and Females of childbearing potential must have agreed to utilize highly effective contraception methods (two separate forms of contraception, one of which must be an effective barrier method, or be nonheterosexually active, practice sexual abstinence, or have a vasectomized partner) from screening throughout the duration of the study period and for 60 days following the last dose of study drug.
* Age ≥ 18 years
* Life expectancy ≥ 1 year

Exclusion Criteria:

* A new AIDS-defining condition diagnosed within 21 days prior to screening
* Females who were breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Proven or suspected acute hepatitis in the 21 days prior to study entry
* Subjects receiving drug treatment for Hepatitis C, or subjects anticipated to receive treatment for Hepatitis C during the course of the study, or with a history of liver disease
* Was experiencing decompensated cirrhosis
* Implanted defibrillator or pacemaker
* Current alcohol or substance abuse judged by the Investigator to potentially interfere with subject compliance
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections requiring parenteral antibiotic or antifungal therapy within 21 days prior to Baseline
* All investigational drugs
* Ongoing therapy or anticipated need to initiate drugs or herbal/natural supplements during the study that were contraindicated or not recommended for use as indicated in the protocol, including drugs not to be used with FTC, RPV, and TDF; or subjects with known allergies to the excipients of the FTC/RPV/TDF STR
* Participation in any other clinical trial without prior approval from the sponsor was prohibited while participating in this trial
* Treatment with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents or systemic steroids during the study (eg, corticosteroids, immunoglobulins, and other immune- or cytokine-based therapies)
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pugatch, MD, Study Director — Gilead Sciences
Locations (18):
- United States (18):
  - Living Hope Clinical Foundation, Long Beach, California
  - Peter J. Ruane MD Inc, Los Angeles, California
  - Anthony Mills MD, Inc., Los Angeles, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Dupont Circle Physicians Group, P.C., Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - The Kinder Medical Group, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Atlanta ID Group, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Northstar Medical Center, Chicago, Illinois
  - Community Research Initiative of New England, Boston, Massachusetts
  - Be Well Medical Center, P.C., Berkley, Michigan
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Southwest Infectious Disease Clinical Research, Inc., Addison, Texas
  - Central Texas Clinical Research, Austin, Texas
  - Peter Shalit, M.D., Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 18 sites in the United States. The first participant was screened on 27 January 2011. The last participant observation was on 26 June 2012.
Pre-assignment Details: 63 participants were screened, 50 were enrolled; 49 participants were treated, and comprise the Safety Analysis set. Participants in the Safety Analysis Set who had no major protocol violation comprise the Full Analysis Set.
Groups:
- FTC/RPV/TDF: Participants switched from their existing treatment regimen of efavirenz (EFV)/emtricitabine (FTC)/tenofovir disoproxil fumarate (tenofovir DF; TDF) to the FTC 200 mg/rilpivirine (RPV) 25 mg/TDF 300 mg single-table regimen (STR).
Period: Overall Study
Arm/Group | FTC/RPV/TDF
Started | 50
Enrolled and Treated | 49
Week 12 (Primary Endpoint) | 49
Completed | 48
Not Completed | 2
Not completed — Enrolled but not treated | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who enrolled and received at least one dose of study drug
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 40
  Black or African American | 6
  Asian | 3
Baseline HIV-1 RNA Category [Number; unit: participants]
  < 50 Copies/mL | 47
  50 to < 400 Copies/mL | 2
EFV plasma concentration [Mean (Standard Deviation); unit: ng/mL] | 2204.9 (1059.42)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 12 (FDA Snapshot Analysis)
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 12 was analyzed using the FDA snapshot analysis.
Time Frame: Week 12
Population: Full Analysis Set: participants who were enrolled into the study, received at least one dose of study drug and had no major protocol violation
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 49
percentage of participants | 100

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 (FDA Snapshot Analysis)
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the FDA snapshot analysis.
Time Frame: Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 49
percentage of participants | 100

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 (FDA Snapshot Analysis)
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the FDA snapshot analysis.
Time Frame: Week 48
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 49
percentage of participants | 93.9

4. Secondary Outcome: Plasma Concentration of RPV and EFV at Week 1
Description: The mean (SD) plasma concentration (ng/mL) of RPV and EFV was measured at Week 1.
Time Frame: Week 1
Population: Participants with evaluable measurements for plasma concentrations of RPV and EFV at Week 1 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 21
ng/mL
  RPV | 31.6 (11.46)
  EFV | 234.5 (234.09)

5. Secondary Outcome: Plasma Concentration of RPV and EFV at Week 2
Description: The mean (SD) plasma concentration (ng/mL) of RPV and EFV was measured at Week 2.
Time Frame: Week 2
Population: Participants with evaluable measurements for plasma concentrations of RPV and EFV at Week 2 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 26
ng/mL
  RPV | 52.3 (24.46)
  EFV | 78.5 (86.91)

6. Secondary Outcome: Plasma Concentration of RPV and EFV at Week 4
Description: The mean (SD) plasma concentration (ng/mL) of RPV and EFV was measured at Week 4.
Time Frame: Week 4
Population: Participants with evaluable measurements for plasma concentrations of RPV and EFV at Week 4 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 27
ng/mL
  RPV | 65.5 (33.19)
  EFV | 10.0 (17.97)

7. Secondary Outcome: Plasma Concentration of RPV and EFV at Week 6
Description: The mean (SD) plasma concentration (ng/mL) of RPV and EFV was measured at Week 6.
Time Frame: Week 6
Population: Participants with evaluable measurements for plasma concentrations of RPV and EFV at Week 6 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 27
ng/mL
  RPV | 67.8 (36.12)
  EFV | 1.9 (4.66)

8. Secondary Outcome: Plasma Concentration of RPV and EFV at Week 8
Description: The mean (SD) plasma concentration (ng/mL) of RPV and EFV was measured at Week 8.
Time Frame: Week 8
Population: Participants with evaluable measurements for plasma concentration of RPV and EFV at Week 8 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 28
ng/mL
  RPV | 76.0 (35.80)
  EFV | NA (NA) — Values were below the limit of quantitation.

9. Secondary Outcome: Plasma Concentration of RPV at Week 12
Description: The mean (SD) plasma concentration (ng/mL) of RPV was measured at Week 12.
Time Frame: Week 12
Population: Participants with measurements for plasma concentration of RPV at Week 12 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 25
ng/mL | 89.0 (54.13)

10. Secondary Outcome: Plasma Concentration of EFV at Week 12
Description: The mean (SD) plasma concentration (ng/mL) of EFV was measured at Week 12. No analyses of EFV plasma concentrations were conducted after Week 12
Time Frame: Week 12
Population: Participants with evaluable measurements for plasma concentration of EFV at Week 12 were analyzed.
Measure: Mean (Inter-Quartile Range); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 17
ng/mL | 45.2 (186.46) [NA to NA] — Interquartile range values were below the limit of quantitation.

11. Secondary Outcome: Plasma Concentration of RPV at Week 24
Description: The mean (SD) plasma concentration (ng/mL) of RPV was measured at Week 24.
Time Frame: Week 24
Population: Participants with evaluable measurements for plasma concentration of RPV at Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 23
ng/mL | 74.1 (37.99)

12. Secondary Outcome: Plasma Concentration of RPV at Week 36
Description: The mean (SD) plasma concentration (ng/mL) of RPV was measured at Week 36.
Time Frame: Week 36
Population: Participants with evaluable measurements for plasma concentration of RPV at Week 36 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 18
ng/mL | 85.5 (34.31)

13. Secondary Outcome: Plasma Concentration of RPV at Week 48
Description: The mean (SD) plasma concentration (ng/mL) of RPV was measured at Week 48.
Time Frame: Week 48
Population: Participants with evaluable measurements for plasma concentration of RPV at Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 24
ng/mL | 77.6 (34.83)

ADVERSE EVENTS:
Time Frame: Baseline to Week 48
Arm/Group | FTC/RPV/TDF
Serious Adverse Events (participants affected / at risk) | 1/49
Other Adverse Events (participants affected / at risk) | 32/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TDF (N=49)
Bradycardia (Cardiac disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TDF (N=49)
Diarrhoea (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 4
Syphilis (Infections and infestations) | 3
Urethritis (Infections and infestations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Insomnia (Psychiatric disorders) | 6
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years